CLINICAL TRIAL: NCT04371991
Title: Can Kisspeptin be Used for Differential Diagnosis of Early Pregnancies?
Brief Title: Kisspeptin Levels in Early Pregnancy
Status: Completed | Type: Observational
Sponsor: Semra Yuksel (Other Government)
Responsible Party: Sponsor-Investigator, Semra Yuksel, Principal investigator, MD, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Other Study IDs: GaziosmanpasaTREH20
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Early Pregnancy; Ectopic Pregnancy
Keywords: kisspeptin; ectopic pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Kisspeptin is a family of peptide hormones encoded by the KISS1 gene. Kisspeptin acts centrally via the kisspeptin receptor to stimulate the release of gonadotropin-releasing hormone (GnRH) from the hypothalamus and has a critical role in the initiation of puberty. Kisspeptin was first discovered as an inhibitor of tumor metastasis and, as a result, was previously known as metastatin. Kisspeptin is also found in high levels in first-trimester syncytiotrophoblast cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Ectopic pregnancy
  Interventions: Diagnostic Test: blood test
- Group 2: Early viable pregnancy
  Interventions: Diagnostic Test: blood test
- Group 3: incomplete miscarriage
  Interventions: Diagnostic Test: blood test
- Group 4: Healthy women
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — blood test (serum samples) for biochemical examination

SUMMARY:
Kisspeptins are a family of neuropeptides that are critical for the puberty initiation and female fertility. The investigators aimed to investigate in this study kisspeptin levels in early pregnancy, ectopic pregnancy, and early pregnancy loss.

DETAILED DESCRIPTION:
Clinicians can easily do a differential diagnosis of early pregnancy, miscarriage, and ectopic pregnancy when the human chorionic gonadotropin (hCG) values higher than 2000 mIU/mL with transvaginal ultrasound. However, in cases where the hCG value is below the critical threshold of 1500 to 2000 mIU/mL (often called the discrimination level) and ultrasound is not likely to be diagnostic, the pregnancy is of unknown location. Plasma or serum kisspeptin is mainly derived from the placenta during pregnancy and plasma kisspeptin levels significantly increase across pregnancy. Plasma kisspeptin levels could be used as a potential biomarker for the discrimination of miscarriage and ectopic pregnancy.

All statistics will be carried out with the use of SPSS (ver. 21, IBM). A P value of <.05 is considered to be statistically significant. Pearson chi-square test will be used to evaluate between-group differences by pregnancy outcome for categoric data. Kisspeptin differences will be calculated between groups with one way ANOVA.

ELIGIBILITY:
Inclusion Criteria:

Women aged between 18-37 years presented with between 5-6 weeks of gestation by last menstrual period.

Exclusion Criteria:

* Women older than 37 years or younger than 18 years
* Women with a molar pregnancy, multiple gestations, gestational age past 6 weeks at the time of blood draw, or if pregnancies were assisted conceptions

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women were considered for the study if they presented between 5-6 weeks of gestation by last menstrual period. Patients were included if they had either confirmed intrauterine pregnancy (IUP) by ultrasound (n=22) or confirmed miscarriage (SAB) by ultrasound (n=20) or ectopic pregnancy.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Kisspeptin levels in early pregnancy | January 2019-January 2020
  Kisspeptin levels can be used for discrimination between ectopic pregnancy and incomplete miscarriage.

CONTACTS AND LOCATIONS:
Overall Officials: sibel bektas, proffessor, Study Chair — Gaziosmanpasa Taksim Education and Research Hospital
Locations (1):
- Gaziosmanpasa Taksim Education and Research Hospital, Istanbul, Turkey (Türkiye)